CLINICAL TRIAL: NCT05620589
Title: The Effect of Different Time Intervals on Rescue Treatment of Helicobacter Pylori Infection: a Prospective, Multicenter Observational Study
Brief Title: The Effect of Time Intervals for Rescue Treatment on Eradication Effect of Helicobacter Pylori Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: Peking University Care Luzhong Hospital (Other); Yuncheng Traditional Chinese Medicine Hospital (Other); Taierzhuang District People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Zibo Central Hospital (Other Government)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Other Study IDs: 2022-SDU-QILU-G006
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Amoxicillin; Tetracycline; Bismuth; Esomeprazole; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; tegoprazan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Amoxicillin + Tetracycline + Bismuth + Esomeprazole: Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Esomeprazole 40mg bid or Amoxicillin 1000mg bid+ Tetracycline 500mg tid+ Bismuth + Esomeprazole 40mg bid
  Interventions: Drug: Amoxicillin + Tetracycline + Bismuth + Esomeprazole
- Amoxicillin + Tetracycline + Bismuth + Vonoprazan: Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth +Vonoprazan 20mg bid or Amoxicillin 1000mg bid+ Tetracycline 500mg tid+ Bismuth + Vonoprazan 20mg bid
  Interventions: Drug: Amoxicillin + Tetracycline + Bismuth + Vonoprazan
- Amoxicillin + Tetracycline 5+ Bismuth + Tegoprazan: Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Tegoprazan 50mg bid or Amoxicillin 1000mg bid+ Tetracycline 500mg tid+ Bismuth + Tegoprazan 50mg bid
  Interventions: Drug: Amoxicillin + Tetracycline + Bismuth + Tegoprazan

INTERVENTIONS:
Drug: Amoxicillin + Tetracycline + Bismuth + Esomeprazole — Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Esomeprazole 40mg bid or Amoxicillin 1000mg bid+ Tetracycline 500mg tid+ Bismuth + Esomeprazole 40mg bid
  Groups: Amoxicillin + Tetracycline + Bismuth + Esomeprazole
Drug: Amoxicillin + Tetracycline + Bismuth + Vonoprazan — Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth +Vonoprazan 20mg bid or Amoxicillin1000mg bid+ Tetracycline 500mg tid+ Bismuth + Vonoprazan 20mg bid
  Groups: Amoxicillin + Tetracycline + Bismuth + Vonoprazan
Drug: Amoxicillin + Tetracycline + Bismuth + Tegoprazan — Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Tegoprazan 50mg bid or Amoxicillin 1000mg bid+ Tetracycline 500mg tid+ Bismuth + Tegopraza 50mg bid
  Groups: Amoxicillin + Tetracycline 5+ Bismuth + Tegoprazan

SUMMARY:
The researchers collect patients who accepted eradication program of the helicobacter pylori but failed to eradicate helicobacter pylor from the outpatient clinic. After rescue therapy, evaluating the effect of retreatment interval on eradication effect of Helicobacter pylori infection.

DETAILED DESCRIPTION:
The researchers collect patients who accepted eradication program of the helicobacter pylori but failed to eradicate helicobacter pylor from the outpatient clinic. Record the interval between the last eradication therapy and this time，6-8 weeks after treatment, the subjects will re-take the 13C-urea breath test. Calculating the eradication rates, adverse reaction rates, patient compliance of each group. Evaluating the effect of retreatment interval on eradication effect of Helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70. Patients with H.pylori infection (Positive for any of the following: 13C/14C-urea breath test, histopathology test, rapid urease test, stool H.pylori antigen test).

Patients who have previously received helicobacter pylori eradication therapy and failed.

Exclusion Criteria:

* Patients with serious underlying diseases, such as liver insufficiency (Aspartate aminotransferase or alanine aminotransferase greater than 1.5 times the normal value), renal insufficiency (Cr≥2.0mg/dL or glomerular filtration rate <50 ml/min), immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%.

Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial.

Patients with active gastrointestinal bleeding. Patients with a history of upper gastrointestinal surgery. Patients allergic to treatment drugs. Patients with medication history of bismuth agents, antibiotics, proton pump inhibitor and other drugs within 4 weeks Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse Patients who are unwilling or incapable to provide informed consents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients in Shandong province,aged between 18 and 70 years old, with positive H. pylori infection that was eradicated by previous therapies but failed are included.
Sampling Method: Probability Sample
Enrollment: 626 (Estimated)
Dates: Start 2022-11-11 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate at different time intervals | immediately after the procedure
  Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Type、Rate and severtiry of adverse reactions | Immediately after the procedure
  Type、Rate and severtiry of adverse reactions
Patient compliance | Immediately after the procedure
  Good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Du LJ, Chen BR, Kim JJ, Kim S, Shen JH, Dai N. Helicobacter pylori eradication therapy for functional dyspepsia: Systematic review and meta-analysis. World J Gastroenterol. 2016 Mar 28;22(12):3486-95. doi: 10.3748/wjg.v22.i12.3486. PMID 27022230
- [Background] Alba C, Blanco A, Alarcon T. Antibiotic resistance in Helicobacter pylori. Curr Opin Infect Dis. 2017 Oct;30(5):489-497. doi: 10.1097/QCO.0000000000000396. PMID 28704226
- [Background] Donelli G, Matarrese P, Fiorentini C, Dainelli B, Taraborelli T, Di Campli E, Di Bartolomeo S, Cellini L. The effect of oxygen on the growth and cell morphology of Helicobacter pylori. FEMS Microbiol Lett. 1998 Nov 1;168(1):9-15. doi: 10.1111/j.1574-6968.1998.tb13248.x. PMID 9812358
- [Background] Catrenich CE, Makin KM. Characterization of the morphologic conversion of Helicobacter pylori from bacillary to coccoid forms. Scand J Gastroenterol Suppl. 1991;181:58-64. PMID 1866596
- [Background] Benaissa M, Babin P, Quellard N, Pezennec L, Cenatiempo Y, Fauchere JL. Changes in Helicobacter pylori ultrastructure and antigens during conversion from the bacillary to the coccoid form. Infect Immun. 1996 Jun;64(6):2331-5. doi: 10.1128/iai.64.6.2331-2335.1996. PMID 8675345
- [Background] Xu HS, Roberts N, Singleton FL, Attwell RW, Grimes DJ, Colwell RR. Survival and viability of nonculturableEscherichia coli andVibrio cholerae in the estuarine and marine environment. Microb Ecol. 1982 Dec;8(4):313-23. doi: 10.1007/BF02010671. PMID 24226049
- [Background] Su X, Chen X, Hu J, Shen C, Ding L. Exploring the potential environmental functions of viable but non-culturable bacteria. World J Microbiol Biotechnol. 2013 Dec;29(12):2213-8. doi: 10.1007/s11274-013-1390-5. Epub 2013 Jun 4. PMID 23733177
- [Background] Lleo MM, Bonato B, Tafi MC, Signoretto C, Boaretti M, Canepari P. Resuscitation rate in different enterococcal species in the viable but non-culturable state. J Appl Microbiol. 2001 Dec;91(6):1095-102. doi: 10.1046/j.1365-2672.2001.01476.x. PMID 11851818
- [Background] Senoh M, Ghosh-Banerjee J, Ramamurthy T, Colwell RR, Miyoshi S, Nair GB, Takeda Y. Conversion of viable but nonculturable enteric bacteria to culturable by co-culture with eukaryotic cells. Microbiol Immunol. 2012 May;56(5):342-5. doi: 10.1111/j.1348-0421.2012.00440.x. PMID 22537150
- [Background] Ozbek A, Ozbek E, Dursun H, Kalkan Y, Demirci T. Can Helicobacter pylori invade human gastric mucosa?: an in vivo study using electron microscopy, immunohistochemical methods, and real-time polymerase chain reaction. J Clin Gastroenterol. 2010 Jul;44(6):416-22. doi: 10.1097/MCG.0b013e3181c21c69. PMID 19904218
- [Background] Liu WZ, Xie Y, Lu H, Cheng H, Zeng ZR, Zhou LY, Chen Y, Wang JB, Du YQ, Lu NH; Chinese Society of Gastroenterology, Chinese Study Group on Helicobacter pylori and Peptic Ulcer. Fifth Chinese National Consensus Report on the management of Helicobacter pylori infection. Helicobacter. 2018 Apr;23(2):e12475. doi: 10.1111/hel.12475. Epub 2018 Mar 7. PMID 29512258
- [Background] Hwang JJ, Lee DH, Lee AR, Yoon H, Shin CM, Park YS, Kim N. Fourteen- vs seven-day bismuth-based quadruple therapy for second-line Helicobacter pylori eradication. World J Gastroenterol. 2015 Jul 14;21(26):8132-9. doi: 10.3748/wjg.v21.i26.8132. PMID 26185386
- [Background] Nyssen OP, Perez-Aisa A, Rodrigo L, Castro M, Mata Romero P, Ortuno J, Barrio J, Huguet JM, Modollel I, Alcaide N, Lucendo A, Calvet X, Perona M, Gomez B, Gomez Rodriguez BJ, Varela P, Jimenez-Moreno M, Dominguez-Cajal M, Pozzati L, Burgos D, Bujanda L, Hinojosa J, Molina-Infante J, Di Maira T, Ferrer L, Fernandez-Salazar L, Figuerola A, Tito L, de la Coba C, Gomez-Camarero J, Fernandez N, Caldas M, Garre A, Resina E, Puig I, O'Morain C, Megraud F, Gisbert JP. Bismuth quadruple regimen with tetracycline or doxycycline versus three-in-one single capsule as third-line rescue therapy for Helicobacter pylori infection: Spanish data of the European Helicobacter pylori Registry (Hp-EuReg). Helicobacter. 2020 Oct;25(5):e12722. doi: 10.1111/hel.12722. Epub 2020 Jul 13. PMID 32656898
- [Background] Fiorini G, Saracino IM, Zullo A, Gatta L, Pavoni M, Vaira D. Rescue therapy with bismuth quadruple regimen in patients with Helicobacter pylori -resistant strains. Helicobacter. 2017 Dec;22(6). doi: 10.1111/hel.12448. Epub 2017 Nov 1. PMID 29094477
- [Background] Lee JW, Kim N, Nam RH, Lee SM, Soo In C, Kim JM, Lee DH. Risk factors of rescue bismuth quadruple therapy failure for Helicobacter pylori eradication. J Gastroenterol Hepatol. 2019 Apr;34(4):666-672. doi: 10.1111/jgh.14625. Epub 2019 Feb 25. PMID 30726563